CLINICAL TRIAL: NCT02578628
Title: Discontinuation of Automated Engagement Support
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data source became unavailable
Sponsor: University of Vermont (Other)
Collaborators: Patient Engagement Systems (Industry); Empire Physicians Medical Group (Other)
Responsible Party: Principal Investigator, Benjamin Littenberg, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 15-453
Record Dates: First submitted 2015-10-10; First posted 2015-10-19 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): These subjects will continue to receive Patient Engagement services.
  Interventions: Other: Patient Engagement
- Control (No Intervention): These patients will have all Patient Engagement services discontinued.

INTERVENTIONS:
Other: Patient Engagement — The patient engagement system monitors routine clinical laboratory test results and sends messages to patients and providers when action is indicated, such as when tests are overdue or results require extra clinical attention. Patients receive first class letters directing them to call their provider. Providers receive fax or electronic messages directing them to reach out to the patient to arrange follow-up care.
  Arms: Active

SUMMARY:
The Chronic Kidney Disease Engagement System is currently in place for 1700 adults receiving care from Empire Physicians Medical Group (EPMG), an Independent Practice Association located in Palm Desert, California. The system monitors routine clinical laboratory test results and send messages to patients and providers when action is indicated, such as when tests are overdue or results require extra clinical attention. This study will assess what happens to laboratory results, utilization of laboratory tests, and costs of care when ther system is discontinued.

DETAILED DESCRIPTION:
The Chronic Kidney Disease Engagement System is currently in place for 1700 adults receiving care from Empire Physicians Medical Group (EPMG), an Independent Practice Association located in Palm Desert, California. The system monitors routine clinical laboratory test results and send messages to patients and providers when action is indicated, such as when tests are overdue or results require extra clinical attention. Patients receive first class letters directing them to call their provider. Providers receive fax or electronic messages directing them to reach out to the patient to arrange follow-up care. It has been used for over three years and appears to have improved adherence to Chronic Kidney Disease (CKD) treatment guidelines by influencing both patient and provider actions. EPMG wishes to restrict the service to those patients with advanced CKD and discontinue it for CKD stages 1-3. The investigators propose implementing this new policy in a randomized fashion with one half of the current early stage patients continuing to receive the service while the other half will no longer receive messages. The investigators will monitor laboratory results and health care utilization for both groups to determine what effect, if any, discontinuation has on quality of care.

Human subjects will either continue to receive letters from the service when their tests are overdue or require additional clinical attention, or will no longer receive the service. All subjects will continue to receive care from their providers. The main outcomes include the frequency of recommended tests for CKD, the level of those tests, and utilization of health care services as indicated by claims data provided by EPMG. No additional data collection will occur beyond that which has been routinely done for clinical care. The study will continue for 36 months.

ELIGIBILITY:
Inclusion Criteria:

Receiving services from Patient Engagement Services at randomization. CKD Stages 1, 2 or 3. Under the care of Empire Physicians Medical Group of Palm Desert, California.

Exclusion Criteria:

Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Claims paid in past 12 months for covered services | 3 years
  Total and breakdown by categories

SECONDARY OUTCOMES:
Lipid test completed within time allotted per disease stage | 3 years
Estimated glomerular filtration | 3 years
Hemoglobin test completed within time allotted per disease stage | 3 years
Serum calcium test completed within time allotted per disease stage | 3 years
Serum phosphorus test completed within time allotted per disease stage | 3 years
Urine albumin-to-creatinine ratio test completed within time allotted per disease stage | 3 years
Serum parathyroid hormone test completed within time allotted per disease stage | 3 years
Serum albumin test completed within time allotted per disease stage | 3 years
Serum electrolytes test completed within time allotted per disease stage | 3 years
Latest LDL <100 mg/dl AND completed within time allotted per disease stage | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Littenberg, MD, Principal Investigator — University of Vermont
Locations (1):
- Empire Physicians Medical Group, Palm Desert, California, United States